CLINICAL TRIAL: NCT00935701
Title: Investigating the Use of Acupressure and Acupuncture With Children With Autism II
Brief Title: Acupressure and Acupuncture as an Intervention With Children With Autism II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Autism Speaks (Other)
Responsible Party: Principal Investigator, Lana Warren, FAC SRVP INSTRUCTOR, Johns Hopkins University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00026158; 2949
Record Dates: First submitted 2009-07-08; First posted 2009-07-09 (Estimated); Results first posted 2014-09-26 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-03

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; Acupressure; Acupuncture
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Acupressure; Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acupuncture and Acupressure (Experimental): In Phase 1, 10 children with ASD will receive acupressure for four weeks. At week 5, they will be introduced to acupuncture which will be continued throughout the rest of the study as tolerated. In Phase 2, 40 children with ASD will receive acupressure twice weekly for 12 weeks. Parents will be trained in the acupressure techniques and will be asked to do this daily, at bedtime, and/or as requested by the child or deemed needed by the parent. Children will begin to be assessed for their ability to participate in acupuncture treatment between weeks 5 and 7 at the discretion of the acupuncturist. By week 7, all children will have been introduced to acupuncture/needling. If needling is still refused at this time, acupressure will continue for the remainder of the study.
  Interventions: Device: Acupressure and Acupuncture

INTERVENTIONS:
Device: Acupressure and Acupuncture — Acupressure involves the stimulation of specific acupoints by firm pressure, while acupuncture involves the insertion of very fine needles (the size of a strand of hair). The needles may be quickly inserted and removed or left in up to 5 minutes at a time.

SUMMARY:
The purpose of this study is to see if children with autism spectrum disorder (ASD) will tolerate an acupressure and acupuncture intervention twice weekly over a 3 month period of time that targets regulatory and behavioral functions. It is anticipated that: 1) children with ASD will tolerate acupressure and, when properly prepared, acupuncture; 2) parents and children will attend bi-weekly appointments over a 3 month period; 3) parents will find administered acupressure technique beneficial to their child and the parent/child relationship; 4) parents will report lower levels of stress regarding their parenting experience. In addition, we will learn information about specific child regulatory and behavior functions (including sleep and attention) from parent and teacher reports while the child receives acupressure and/or acupuncture. A small clinical trial will be conducted with 50 eligible children (3-10 years of age) with ASD (and one parent each) who will be enrolled into two groups: Phase 1 pre-pilot group of 10 children who will complete 8 weeks of treatment to help develop a treatment protocol; Phase 2 with 40 children treated for 12 weeks. Parents and teachers will complete pre-intern and post surveys, and children who do not tolerate acupressure/acupuncture will be counted as "treatment failures" for analyses.

DETAILED DESCRIPTION:
This study will be conducted in two phases. In Phase 1, we will have 10 children with ASD (and 1 parent each for each child). The children will receive acupressure for four weeks. At week five, they will be introduced to acupuncture which will be continued throughout the rest of the study as tolerated. Sessions will be twice weekly and 30 minutes in length with the exception of the first session which will include an assessment and treatment session and be approximately an hour and a half. The total study period for Phase 1 is 8 weeks. The study acupuncturist has developed a proposed treatment protocol for children with ASD based upon the works cited above and his own clinical experience. This will be further developed and refined during the Phase I portion of this research. During the first session, which will include a TCM assessment and an initial treatment session, the acupuncturist will determine and initiate a treatment approach utilizing the 7 meridians and 4 points listed below based upon the assessment findings. Order of the treatment and direction of the strokes will be at the discretion of the acupuncturist. When treatment is introduced, this will be demonstrated, if deemed necessary by the practitioner, on a doll, the clinician or parent. Treatment involves points and pathways located on the child's arms, hands, feet and legs only. It will include:

1. Meridians: Acupressure to the following meridians until acupuncture is introduced ( these are also the strokes the parents will use at home throughout the duration of the treatment phase of the study):

   1. Heart (arm)
   2. Spleen (leg)
   3. Stomach (leg)
   4. Kidney (leg)
   5. Bladder (leg)
   6. Liver (leg)
   7. Gallbladder (leg)
2. Points: Focus on the following points throughout the study period:

   1. Ht 7 (arm)
   2. St 36 (leg)
   3. SP 6 (leg)
   4. Ki 3 (leg)
3. Additional Points: After the initial 4 weeks of acupressure reassess the child and begin, as tolerated, to introduce acupuncture treatment from the same acupuncture point list as identified above as well as the following extra points related specifically to the individual child's condition.

Ht 8 Clears heat from the heart (hand) Liv 2 Clears heat from the body (foot) Liv 3 Calms mind and body and diffuses emotions (foot) St 41 Clears heat (foot) St 44 Clears heat from the body (foot) Sp 4 Tonifies spleen Qi (foot) GB 41 Clears heat (leg) GB 43 Hot phlegm (foot)

From our experience with these children in Phase I, we will create a preliminary manual with guidelines for introducing acupressure to children with ASD, for transitioning to acupuncture, and for maintaining continued participation in the intervention. This manual will be reviewed by the Advisory Committee and occupational therapist for further comment as well as submitted to the IRB before proceeding to Phase 2.

In Phase 2, we will conduct a preliminary clinical trial with 40 eligible children with ASD (and one parent for each child). The children will receive the manualized intervention twice weekly for 12 weeks for a total of up to 24 sessions. As above, sessions will be 30 minutes in length.

Children who refuse or cannot tolerate acupressure by the fourth session will be discontinued from the study and another subject added. Parents will be trained in the acupressure techniques beginning with the first treatment session and will be asked to do this daily, at bedtime, and/or as requested by the child or deemed needed by the parent e.g. if child finds the study procedure calming, parent may initiate if child's behavior is escalating. Depending upon the child's response, this will take up to 15 minutes. Parents will be instructed not to perform acupressure if the child resists, but to continue to offer this each night. When parents are taught the techniques, they will be given an oral explanation with physical demonstration and written instructions with diagram. They will observe, do and teach and will be assessed for their proficiency at performing acupressure by the acupuncture practitioner. This will be done by observing the parent perform the acupressure strokes on the child and assessing pressure, accuracy, direction and speed. Parents will be given a structured diary which will include types of observations to make and minimum frequency.

Children will begin to be assessed for their ability to participate in acupuncture treatment between weeks 5 and 7 at the discretion of the acupuncturist. This will be determined by factors such as the child's receptivity and acceptance to touch during acupressure sessions, willingness to be treated, observation of relaxation during treatment, their reaction to being introduced to the needles, and report of positive behavioral changes by the child and/or parent. The child will be able to see and touch a needle as well as witness an insertion in the arm of the practitioner (or doll or parent) as deemed necessary by the practitioner. The child's reaction to this introduction will determine when the actual needling will begin. Needling will only begin with the child's verbal agreement. By week 7, all children will have been introduced to acupuncture/needling. If needling is still refused at this time, acupressure will continue for the remainder of the study.

Due to potential vacations, illnesses, and other events, the 24 treatments (16 for Phase 1) can occur over a 15 week period (10 for Phase 1), with no more than 2 sessions per week. Each child must participate in a minimum of 75% of the sessions (18 for Phase 2; 12 for Phase 1) to be included in the study. If a child misses sufficient sessions so that he/she is not able to meet the study criteria, treatment will be discontinued at that time.

Children failing to meet this criteria due to unavoidable circumstances (e.g., family vacation, unrelated illness) will not be considered in analyses of study data. All other children failing to meet this criterion will be considered to have failed to tolerate acupuncture. One parent and the child's primary teacher will be asked to fill out questionnaires which will take parents approximately 70-120 minutes to complete and teachers approximately 45-70 minutes to complete on 3 different occasions (before, during and after the treatment). The parent will fill out five questionnaires that address the child's behavior, sleep, and parental level of stress. Questionnaires include: Behavior Assessment Scale for Children, Conners' Rating Scales, PDD Behavior Inventory, Parenting Stress Inventory and the Children's Sleep Inventory. The parent will also complete two additional questionnaires: Autism Parent Survey and Autism Child Survey. These questionnaires are designed to ascertain participants' response to treatment. One questionnaire is for the parent to complete, and the other is for the parent to complete together with the child, if possible. The teacher will fill out the Behavior Assessment Scale for Children, Conners' Rating Scales, and PDD Behavior Inventory,. The parent will sign a letter that is addressed to the teacher from the Primary Investigator that gives the teacher permission to complete the forms. The parent will also be asked to keep a structured diary (provided) noting any changes in behavior that they notice. Entries are to be made at a minimum weekly. The acupuncturist will remind parents to complete these entries each week.

Phase 1 eligibility assessments will be conducted at Kennedy Krieger Institute Center for Autism and Related Disorders (CARD) and acupressure/acupuncture treatment sessions will be conducted at the CARD treatment rooms or at the acupuncturist's Catonsville offices.

Phase 2 will occur in two different locations (Baltimore and Laurel/Silver Spring) at two different times to allow for a larger sample size and to be more convenient to families. At the conclusion of the study, parents will be kept informed of any publications that are the result of this study. Parents may also receive the acupuncturist's notes on the participant if requested.

ELIGIBILITY:
Inclusion Criteria:

* In addition to qualifying by age and IQ (IQ of at least 50), children will meet two of three of the following criteria for ASD (PDD-NOS, Autism or Asperger Syndrome): (1) Autism Diagnostic Observation Schedule-Generic, (ADOS-G) algorithm criteria for ASD or Autism, (Lord, Rutter, DiLavore, & Risi, 2001) (2) Autism Diagnostic Interview-Revised, (ADI-R) algorithm criteria (Lord, Rutter, & Le Couteur, 2003) meeting criteria for autism for the social or communication domain by being within 2 points of the algorithm cut-off for autism on the other, or coming within 1 point of the cut-off for autism on both and (3) have clinical judgment of autism, PDD-NOS or Asperger Syndrome by an autism expert. All of the ADOS-G testing sessions will be videotaped with inter-rater reliability being conducted on 20% of children tested. These videotapes will be destroyed following determination of study eligibility for those found not eligible. For those who are eligible, the videotapes will be destroyed after eligibility is determined or, for the 20% used for determining inter-rater reliability, the videotapes will be destroyed following this analysis. Parents will be asked not to start any new intervention or modification of current intervention during the study period unless deemed absolutely necessary. If such a change has to be made, the parents are requested to inform the Principal Investigator and either participation will be discontinued (without consideration as a treatment failure) or data subsequent to that point will be excluded from analyses.

Exclusion Criteria:

* Children who have had any significant medication or treatment change within the past four weeks prior to the beginning of the study, children who are in foster care, children with a bleeding disorder, children who are not proficient in English, children who do not have normal hearing with or without aides, and children failing to meet inclusion criteria will not be eligible for the study. If a child has a significant change in his entrance treatment program (e.g.; significant change in medication, school placement) during the study, the PI in consultation with Advisory Committee members, Dr. Rebecca Landa and Dr. Andrew Zimmerman, both autism research experts, will determine if the child is appropriate to remain in the study. Parents who are not proficient in English will not be included in the study.

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2009-07; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lana Warren, Ed.D., Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Locations (1):
- Kennedy Krieger Institute, Baltimore, Maryland, United States

REFERENCES:
- [Background] Hanson E, Kalish LA, Bunce E, Curtis C, McDaniel S, Ware J, Petry J. Use of complementary and alternative medicine among children diagnosed with autism spectrum disorder. J Autism Dev Disord. 2007 Apr;37(4):628-36. doi: 10.1007/s10803-006-0192-0. PMID 16977497
- [Background] Green VA, Pituch KA, Itchon J, Choi A, O'Reilly M, Sigafoos J. Internet survey of treatments used by parents of children with autism. Res Dev Disabil. 2006 Jan-Feb;27(1):70-84. doi: 10.1016/j.ridd.2004.12.002. PMID 15919178
- [Background] Flaws, B. (1997) A Handbook of TCM Pediatrics. Michigan: Blue Poppy Press.
- [Background] Clark, E., & Zhou, Z. (2005). Autism in China: From acupuncture to applied behavior analysis. Psychology in the Schools, 42(3), 285-295.
- [Background] Cullen L, Barlow J. 'Kiss, cuddle, squeeze': the experiences and meaning of touch among parents of children with autism attending a Touch Therapy Programme. J Child Health Care. 2002 Sep;6(3):171-81. doi: 10.1177/136749350200600303. PMID 12224834
- [Background] Cullen-Powell LA, Barlow JH, Cushway D. Exploring a massage intervention for parents and their children with autism: the implications for bonding and attachment. J Child Health Care. 2005 Dec;9(4):245-55. doi: 10.1177/1367493505056479. PMID 16275663
- [Background] Escalona A, Field T, Singer-Strunck R, Cullen C, Hartshorn K. Brief report: improvements in the behavior of children with autism following massage therapy. J Autism Dev Disord. 2001 Oct;31(5):513-6. doi: 10.1023/a:1012273110194. PMID 11794416

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Ten children with ASD (8 boys and 2 girls between the ages of 3 and 10 years) and their parents took part in a 16-week intervention. Children were recruited through autism networks and Kennedy Krieger Institute. Phase 2 was not conducted due to difficulty recruiting enough participants to successfully complete a randomized controlled trial.
Pre-assignment Details: All participants completed 16 treatment sessions and all parents carried out a home component of treatment during this time period.
Period: Overall Study
Arm/Group | Acupuncture and Acupressure
Started | 10
Transition Acupressure to Acupuncture | 9
Completed | 9
Not Completed | 1
Not completed — Failure to Transition to Acupuncture | 1

BASELINE CHARACTERISTICS:
Arm/Group | Acupuncture and Acupressure
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.2 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Proportions of Children Completing Acupressure and Acupuncture Treatment.
Time Frame: 2 months into Phase 1
Population: Participants who transitioned from acupressure to acupuncture were assessed.
Measure: Number; unit: participants
Groups:
- Primary Group: Phase 1
Arm/Group | Primary Group
Number analyzed (Participants) | 9
participants | 9

2. Secondary Outcome: Change in Conners' Rating Scales
Description: The Conners' Rating Scales Revised (CRS-R) is used to assess attention deficit hyperactivity disorder (ADHD) as well as other related behavioral concerns. The CRS-R is made up of 14 scales. Analysis was done on 6 of these scales: Conners' Global Index Restless-Impulsive, Conners' Global Index Emotional Lability, Conners' Global Index Total, DSM-IV Inattentive, DSM-IV Hyperactive-Impulsive, and DSM-IV Total. Raw scores are converted to T-scores, based on age and gender of the child. A high T-score indicates a greater number and/or frequency of reported concerns. Pre T-scores were subtracted from post T-scores to calculate the change in T-score.
Time Frame: Pre intervention (baseline), post intervention (8 weeks)
Measure: Mean (Standard Deviation); unit: t-scores
Arm/Group | Primary Group
Number analyzed (Participants) | 9
t-scores
  Restless-Impulsive | -8.67 (8.2)
  Emotional Lability | -5 (8.4)
  Global Index Total | -8.11 (8.49)
  DSM-IV Inattentive | -11.11 (8.58)
  DSM-IV Hyperactive-Impulsive | -8 (9.71)
  DSM-IV Total | -9.78 (9.56)
Statistical Analysis 1: Comparison: Primary Group; Mean change in score from pre to post on Restless-Impulsive subscale; Test type: Superiority or Other; p = 0.01, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Primary Group; Mean change in score from pre to post on Emotional Lability subscale; Test type: Superiority or Other; p = 0.09, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Primary Group; Mean change in score from pre to post on Global Index Total; Test type: Superiority or Other; p = 0.02, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Primary Group; Mean change in score from pre to post on DSM-IV Inattentive subscale; Test type: Superiority or Other; p = 0.01, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Primary Group; Mean change in score from pre to post on DSM-IV Hyperactive-Impulsive subscale; Test type: Superiority or Other; p = 0.03, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Primary Group; Mean change in score from pre to post on DSM-IV Total; Test type: Superiority or Other; p = 0.01, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change in Children's Sleep Habits Questionnaire
Description: The Children's Sleep Habits Questionnaire (CSHQ) assesses sleep problems common in school-age children and is comprised of eight subscales. Each item receives a score from 1 (meaning the problem occurs rarely) to 3 (meaning the problem usually occurs); therefore, a higher score is the worse outcome. Scale ranges are as follows: Bedtime Resistance: 6 to 18, Sleep Onset Delay: 1 to 3, Sleep Duration: 3 to 9, Sleep Anxiety: 4 to 12, Night Wakings: 3 to 9, Parasomnias: 7 to 21, Disordered Breathing: 3 to 9, Daytime Sleepiness: 8 to 24, and Total Disturbance (items from all scales): 33 to 99. Subscale scores from pre intervention were subtracted from post subscale scores in order to get the change in scores.
Time Frame: Pre intervention (baseline), post intervention (8 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Primary Group
Number analyzed (Participants) | 10
units on a scale
  Bedtime Resistance | -.4 (.7)
  Sleep Onset Delay | -.6 (.7)
  Sleep Duration | -.3 (1.25)
  Sleep Anxiety | -.22 (1.09)
  Night Wakings | -.33 (1.66)
  Parasomnias | .56 (1.13)
  Disordered Breathing | 0 (0)
  Daytime Sleepiness | -.78 (1.99)
  Total Disturbance | -2.44 (3.54)
Statistical Analysis 1: Comparison: Primary Group; Mean change in score from pre to post on Bedtime Resistance subscale; Test type: Superiority or Other; p = 0.08, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Primary Group; Mean change in score from pre to post on Sleep Onset Delay subscale; Test type: Superiority or Other; p = 0.03, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Primary Group; Mean change in score from pre to post on Sleep Duration subscale; Test type: Superiority or Other; p = 0.82, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Primary Group; Mean change in score from pre to post on Sleep Anxiety subscale; Test type: Superiority or Other; p = 0.58, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Primary Group; Mean change in score from pre to post on Night Wakings subscale; Test type: Superiority or Other; p = 0.66, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Primary Group; Mean change in score from pre to post on Parasomnias subscale; Test type: Superiority or Other; p = 0.18, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Primary Group; Mean change in score from pre to post on Daytime Sleepiness subscale; Test type: Superiority or Other; p = 0.31, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Primary Group; Mean change in score from pre to post on Total Disturbance; Test type: Superiority or Other; p = 0.07, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Change in Parenting Stress Index
Description: The Parenting Stress Index (PSI) was designed for parents of children ages 1:6 to 12:5 and identifies stressors in the parent-child relationship. Specifically, the PSI measures child's characteristics on six subscales, which are summed get a total score in the child domain (47 to 235). The PSI also has seven subscales that measure parent characteristics, and are summed to get a total score in the parent domain (54 to 270). The totals from the parent and child domains are summed for a total stress score (101 to 505). Higher scores indicate a higher level of stress. Pre scores were subtracted from post scores in order to get the change in scores.
Time Frame: Pre intervention (baseline), post intervention (8 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Primary Group
Number analyzed (Participants) | 10
units on a scale
  Child Domain Total | -11.67 (12.19)
  Parent Domain Total | -4 (10.74)
  Total Stress | -15.67 (19.72)
Statistical Analysis 1: Comparison: Primary Group; Mean change in score from pre to post on Child Domain Total; Test type: Superiority or Other; p = 0.04, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Primary Group; Mean change in score from pre to post on Parent Domain Total; Test type: Superiority or Other; p = 0.31, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Primary Group; Mean change in score from pre to post on Total Stress; Test type: Superiority or Other; p = 0.07, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Description: None of the ten participants experienced serious and/or other [non-serious] adverse events related to this study's protocol.
Arm/Group | Primary Group
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

LIMITATIONS AND CAVEATS:
There were no limitations to this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No